CLINICAL TRIAL: NCT02058329
Title: A Geriatric Home Visit Program to Reduce Post Hip Fracture Morbidity and Mortality
Brief Title: A Geriatric Home Visit Program to Reduce Post-Hip Fracture Complications
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Many patients were lost to follow-up
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Garbis Dabaghian, M.D., Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08-023
Record Dates: First submitted 2012-10-25; First posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Fracture; Infection; Depression; Gait Instability; Debility
Keywords: Hip fracture; postoperative complications; Depression; Environmental Hazards; FIM scores; Falls
MeSH Terms: conditions — Fractures, Bone; Infections; Depression; Gait Disorders, Neurologic; Frailty; Hip Fractures; Postoperative Complications | interventions — House Calls

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention): Standard of care with no home visit
- Home Visit (Experimental): After the post hip-fracture patient is discharged to home, there will be home visits by a geriatric fellow assess overall function and response to treatment/s by depression screen, FIM scores, and environmental risk assessment
  Interventions: Other: Home Visit

INTERVENTIONS:
Other: Home Visit — A geriatric fellow will conduct a comprehensive in hospital post discharge assessment of hip fracture patients discharged to home in the intervention group.Follow up home visits will occur at 1,3 and 6 months post discharge.Any problems will be referred to the patient's primary care physician.
  Arms: Home Visit

SUMMARY:
The overall goal of the project is to reduce the incidence of post hip fracture morbidity and mortality by conducting geriatric fellow periodic home visits.The assessment will be multidisciplinary and will include assessments of functional status, depression, environmental risks and medical conditions. This group will be compared against a group followed by the usual standard of care post hip fracture.

DETAILED DESCRIPTION:
All patients post hip fracture on the hospital's rehabilitation service that will be discharged to home will be enrolled after obtaining consent. Patients will be randomized into the intervention group and the usual standard of care group.We will be recruiting a total of 100 patients , with equal numbers for each group.All patients will undergo an initial assessment by a Geriatric fellow prior to discharge . The intervention group will be seen at the time of discharge in the hospital and at home at 1, 3, and 6 months post hip fracture. The control group will be seen at the time of discharge in the hospital and then again at 6 months for follow up. The two groups will then be compared for multiple known complications post hip fractures well as mortality.

ELIGIBILITY:
Inclusion Criteria:

* All post hip fracture patients on the hospital's rehabilitation service being discharged to home .

Exclusion Criteria:

* Patients discharged to nursing homes or rehabilitation facilities.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Decreased rate of depression, falls, medication errors and post-op-complications | 6 months and 1 year
  geriatric depression screen, FIM score, medication reconciliation

SECONDARY OUTCOMES:
environmental hazards will be identified | 6 months and 1 year
  safety inspection of home

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jarrett, M.D., Principal Investigator — Staten Island University Hospital; Marianne Smith, M.D., Study Director — Staten Island University Hospital; Garbis Dabagian, M.D., Principal Investigator — Staten Island University Hospital; Donna Seminara, M.D., Principal Investigator — Staten Island University Hospital; Jeffery Weinberg, M.D., Principal Investigator — Staten Island University Hospital; Mario Castellanos, M.D., Principal Investigator — Staten Island University Hospital; Anita Szerszen, M.D., Principal Investigator — Staten Island University Hospitial
Locations (1):
- Staten Island University Hospital, Staten Island, New York, United States

REFERENCES:
- [Background] McGinn T, Conte JG, Jarrett MP, ElSayegh D. Decreasing mortality for patients undergoing hip fracture repair surgery. Jt Comm J Qual Patient Saf. 2005 Jun;31(6):304-7. doi: 10.1016/s1553-7250(05)31038-5. PMID 15999957